CLINICAL TRIAL: NCT05221931
Title: Drug-Coated Balloon Versus Drug-Eluting Stent for Treatment of De-Novo Coronary Lesions in Patients With High Bleeding Risk (DCB-HBR Trial)
Brief Title: Drug-Coated Balloon in Patients With High Bleeding Risk
Acronym: DCB-HBR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Seoul National University Bundang Hospital (Other); Korea University Ansan Hospital (Other); Chonnam National University Hospital (Other); Chung-Ang University Gwangmyeong Hospital (Other); Gangneung Asan Hospital, University of Ulsan College of Medicine (Unknown); Gyeongsang National University Hospital (Other); Uijeongbu St. Mary Hospital (Other); Keimyung University Dongsan Medical Center (Other); Inha University Hospital (Other); Chungbuk National University (Other); Wonju Severance Christian Hospital (Other); SMG-SNU Boramae Medical Center (Other); Kangbuk Samsung Hospital, Sungkyunkwan University (Other); Ewha Womans University (Other); Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCBHBR2021-12-111-001
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; De-Novo Coronary Lesion; Drug-Coated Balloon; High Bleeding Risk; Prognosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label, randomized controlled, noninferiority trial
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DES group (Active Comparator): Patients will be randomized to either the DCB group or the DES group with 1:1 ratio during the index procedure after diagnostic angiography.
  In DES group, latest second-generation DES will be used (Ultimaster Tansei) during the index procedure
  Interventions: Procedure: Percutaneous coronary intervention
- DCB group (Experimental): Patients will be randomized to either the DCB group or the DES group with 1:1 ratio during the index procedure after diagnostic angiography.
  In DCB group, Agent (Boston Scientific, USA), Prevail (Medtronic, USA), or SeQuent Please, SeQuent Please NEO (B-Braun, Germany) will be used during the index procedure.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — 1:1 randomization to DES (Ultimaster Tansei) or DCB (Agent [Boston Scientific, USA], Prevail [Medtronic, USA], or SeQuent Please, SeQuent Please NEO [B-Braun, Germany])

SUMMARY:
DCB-HBR trial is prospective, multi-center, open-label, randomized controlled, noninferiority trial.

The aim of the study is to compare clinical outcomes of drug-coated balloon (DCB) with drug-eluting stent (DES) for treatment of de-novo coronary lesion in patients with high bleeding risk (HBR).

DETAILED DESCRIPTION:
Second-generation DES is the standard of care for patients with coronary artery disease who are deemed eligible for percutaneous coronary intervention (PCI). Despite many advantages, DES inevitably accompany disadvantages such as the occurrence of late stent thrombosis and the need for maintaining dual antiplatelet (DAPT) for certain period due to permanent vascular implant, which lead to both increased ischemic and bleeding events.

As an alternative to DES, drug-coated balloon (DCB), a novel treatment strategy, which has benefit of having shorter DAPT maintenance duration due to the absence of metallic scaffolds and polymers, has been introduced. Based on meta-analysis based on many randomized clinical trials (RCT), its use has been established in in-stent restenosis of bare-metal stents (BMS) and DES. Furthermore, recently published RCT demonstrated efficacy and safety of DCB in de-novo coronary lesions in small vessels with reference vessel size<3.0mm. However, studies exploring the feasibility of DCB in de-novo coronary artery stenosis beyond small vessels are limited. Furthermore, there is scarce data comparing DCB with DES in patients with de-novo coronary artery stenosis and high bleeding risk (HBR), a situation in which long-term maintenance of DAPT is a clinical dilemma. In previous BASKET-SMALL 2 trial, DCB showed noninferiority to DES in patients with de-novo coronary artery stenosis and small vessel disease. However, this trial was conducted in non-HBR patients, and the number of participated patients was insufficient. In another RCT, DEBUT trial exclusively enrolled patients with HBR and de-novo coronary artery stenosis. Although the DEBUT trial showed superiority of DCB angioplasty over implantation of BMS to treat de-novo coronary artery stenosis in patients with HBR, the results could not be applicable in contemporary practice because BMS has been no longer in clinical use. Recently, multiple RCTs have proved short-term DAPT (1-3 months) has comparable efficacy to longer term DAPT in HBR patients using latest second-generation DES.

On this background, the current trial aims to compare clinical outcomes between DCB and DES to treat de-novo coronary artery stenosis in patients with HBR receiving guideline-directed short-term DAPT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 19 years of age
2. Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.
3. Patients with at least one lesion with greater than 50% diameter stenosis or fractional flow reserve ≤0.80 requiring revascularization in de-novo coronary artery of reference vessel size ≥2.25 mm
4. Patients with high bleeding risk: one or more of the criteria listed (1) Adjunctive oral anticoagulation treatment planned to continue after PCI (2) Age ≥ 75 years old (3) Baseline Hemoglobin <11 g/dl (or anemia requiring transfusion during the 4 weeks prior to randomization) (4) Any prior intra-cerebral bleeding (5) Stroke at any time or transient ischemic attack in the previous 6 months. (6) Hospital admission for bleeding during the prior 12 months (7) Non skin cancer diagnosed or treated < 3 years (8) Planned daily NSAID (other than aspirin) or steroids for >30 days after PCI (9) Planned surgery that would require interruption of DAPT (within next 12 months) (10) Renal failure defined as calculated creatinine clearance <40 ml/min or on dialysis (11) Hematological disorders (platelet count <100,000/mm3 or any coagulation disorder) (12) Severe chronic liver disease defined as patients who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice (13) Expected non-compliance to prolonged DAPT for other medical reasons

Exclusion Criteria:

1. Patients unable to provide consent
2. Patients with known intolerance to aspirin, P2Y12 inhibitors, or components of drug-eluting stents
3. Patients with angiographic findings of (1) Left main coronary artery disease (2) In-stent restenosis is the cause of target lesion (3) Target lesion in bypass graft (4) True bifurcation lesion that requires upfront 2-stenting
4. Patients who have non-cardiac co-morbid conditions with life expectancy <2 year
5. Patients who may result in protocol non-compliance (site investigator's medical judgment)
6. Patients with cardiogenic shock or cardiac arrest
7. Patients with severe left ventricular systolic dysfunction (ejection fraction <30%)
8. Patients with severe valvular heart disease requiring open heart surgery
9. Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1359 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 2 years from last patient enrollment
  a composite of cardiovascular death, target-vessel myocardial infarction (MI), and clinically indicated target-vessel revascularization (TVR)

SECONDARY OUTCOMES:
BARC type 2, 3 or 5 bleeding (Major secondary endpoint) | 2 years from last patient enrollment
  BARC type 2, 3 or 5 bleeding
Cardiovascular death | 2 years from last patient enrollment
  Cardiovascular death
All-cause death | 2 years from last patient enrollment
  All-cause death
Target-vessel MI | 2 years from last patient enrollment
  Target-vessel MI
Non-target vessel related MI | 2 years from last patient enrollment
  Non-target vessel related MI
Non-fatal MI | 2 years from last patient enrollment
  Non-fatal MI
Clinically indicated target-lesion revascularization (TLR) | 2 years from last patient enrollment
  Clinically indicated target-lesion revascularization (TLR)
Clinically indicated TVR | 2 years from last patient enrollment
  Clinically indicated TVR
Non-target vessel revascularization | 2 years from last patient enrollment
  Non-target vessel revascularization
Any revascularization | 2 years from last patient enrollment
  Any revascularization
Vessel or stent thrombosis | 2 years from last patient enrollment
  definite by Academic Research Consortium (ARC) definition
Cardiovascular death or target-vessel MI | 2 years from last patient enrollment
  Cardiovascular death or target-vessel MI
Target vessel failure without procedure-related MI | 2 years from last patient enrollment
  a composite of cardiovascular death, target-vessel myocardial infarction (MI) without procedure-related MI, and clinically indicated target-vessel revascularization (TVR)
Target lesion failure (TLF) | 2 years from last patient enrollment
  a composite of cardiovascular death, target-vessel MI, and clinically indicated TLR
Cardiovascular death, target-vessel MI, or vessel or stent thrombosis | 2 years from last patient enrollment
  Cardiovascular death, target-vessel MI, or vessel or stent thrombosis
All-cause death, non-fatal MI, or any revascularization | 2 years from last patient enrollment
  All-cause death, non-fatal MI, or any revascularization
Bleeding according to BARC definition | 2 years from last patient enrollment
  Bleeding according to BARC definition
Bleeding according to TIMI definition | 2 years from last patient enrollment
  Bleeding according to TIMI definition
Cerebrovascular accident (CVA) | 2 years from last patient enrollment
  Ischemic stroke, Hemorrhagic stroke, Transient ischemic attack (TIA)
Target vessel failure (TVF) at Extended Follow-up | 4 years from last patient enrollment
  a composite of cardiovascular death, target-vessel myocardial infarction (MI), and clinically indicated target-vessel revascularization (TVR) at Extended Follow-up
BARC type 2, 3 or 5 bleeding (Major secondary endpoint) at Extended Follow-up | 4 years from last patient enrollment
  BARC type 2, 3 or 5 bleeding at Extended Follow-up
Cardiovascular death at Extended Follow-up | 4 years from last patient enrollment
  Cardiovascular death at Extended Follow-up
All-cause death at Extended Follow-up | 4 years from last patient enrollment
  All-cause death at Extended Follow-up
Target-vessel MI at Extended Follow-up | 4 years from last patient enrollment
  Target-vessel MI at Extended Follow-up
Non-target vessel related MI at Extended Follow-up | 4 years from last patient enrollment
  Non-target vessel related MI at Extended Follow-up
Non-fatal MI at Extended Follow-up | 4 years from last patient enrollment
  Non-fatal MI at Extended Follow-up
Clinically indicated target-lesion revascularization (TLR) at Extended Follow-up | 4 years from last patient enrollment
  Clinically indicated target-lesion revascularization (TLR) at Extended Follow-up
Clinically indicated TVR at Extended Follow-up | 4 years from last patient enrollment
  Clinically indicated TVR at Extended Follow-up
Non-target vessel revascularization at Extended Follow-up | 4 years from last patient enrollment
  Non-target vessel revascularization at Extended Follow-up
Any revascularization at Extended Follow-up | 4 years from last patient enrollment
  Any revascularization at Extended Follow-up
Vessel or stent thrombosis at Extended Follow-up | 4 years from last patient enrollment
  definite ㅍessel or stent thrombosis at Extended Follow-up by Academic Research Consortium (ARC) definition
Target vessel failure without procedure-related MI at Extended Follow-up | 4 years from last patient enrollment
  a composite of cardiovascular death, target-vessel myocardial infarction (MI) without procedure-related MI, and clinically indicated target-vessel revascularization (TVR)
Cardiovascular death or target-vessel MI at Extended Follow-up | 4 years from last patient enrollment
  Cardiovascular death or target-vessel MI at Extended Follow-up
Target lesion failure (TLF) at Extended Follow-up | 4 years from last patient enrollment
  Target lesion failure (TLF) at Extended Follow-up
Cardiovascular death, target-vessel MI, or vessel or stent thrombosis at Extended Follow-up | 4 years from last patient enrollment
  Cardiovascular death, target-vessel MI, or vessel or stent thrombosis at Extended Follow-up
All-cause death, non-fatal MI, or any revascularization at Extended Follow-up | 4 years from last patient enrollment
  All-cause death, non-fatal MI, or any revascularization at Extended Follow-up
Bleeding according to BARC definition at Extended Follow-up | 4 years from last patient enrollment
  Bleeding according to BARC definition at Extended Follow-up
Bleeding according to TIMI definition at Extended Follow-up | 4 years from last patient enrollment
  Bleeding according to TIMI definition at Extended Follow-up
Cerebrovascular accident (CVA) at Extended Follow-up | 4 years from last patient enrollment
  Ischemic stroke, Hemorrhagic stroke, Transient ischemic attack (TIA)

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (17):
- South Korea (17):
  - Korea University Ansan Hospital, Ansan
  - Chungbuk National University, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - Gangneung Asan Hospital, University of Ulsan College of Medicine, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Inha University Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Ewha Womans University College of Medicine, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Kuro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Supporting Information: Study Protocol, CSR
Time Frame: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked